CLINICAL TRIAL: NCT06166290
Title: CO2 LASER Vaporization vs Electrosurgical Fulguration for the Surgical Management of Perianal Condyloma: a Randomized Controlled Trial.
Brief Title: Comparing CO2 Laser and Electrosurgical Treatments for Perianal Condyloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Gerald Gantt, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY2023-1221
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Perianal Wart

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CO2 LASER Vaporization Group (Experimental)
  Interventions: Procedure: CO2 LASER Vaporisation
- Electrosurgical Fulguration Group (Active Comparator)
  Interventions: Procedure: Electrosurgical Fulguration

INTERVENTIONS:
Procedure: CO2 LASER Vaporisation — The CO2 LASER vaporization procedure is described as follows. Patient positioning will be done, and patient will be anesthetized. Local infiltration with 2% lidocaine, nerve block or general anesthesia will be given. The surgical field will be disinfected and draped. The perianal and anal area will be investigated for lesion. CO2 LASER from 20 cm distance in a continuous wave mode and 20 W power will be applied. After warts melts, necrotic tissue will be removed. After the operation was completed, residual debris will be wiped away with a piece of moist gauze. Bacitracin cream applied over the treated areas. Upon discharge acetaminophen 1-gram q8 and Ibuprofen 600 q8 for pain.
  Arms: CO2 LASER Vaporization Group
Procedure: Electrosurgical Fulguration — The procedure is described as follows. Patient will be administered regional or general anesthesia, placed in prone jack-knife position. Prepping and draping will be done. The perianal and anal area will be investigated for lesion. The lesions will be excised, and the bases will be fulgurated. Electrosurgery device will be used in monopolar setting (30 Cut mode, 30 Coag mode). After procedure local analgesics total MERCAINE/EPI 0.25% 20 ml on both sides of the lesion. Bacitracin cream applied over the treated areas. Upon discharge 1000 mg of Tylenol every 8 hours along with 600 mg of ibuprofen every 8 hours.
  Arms: Electrosurgical Fulguration Group

SUMMARY:
Perianal condyloma are skin- colored and fleshy lesions caused by various variants of Human Papilloma Virus (HPV), most commonly 6 and 11. The treatment modalities available include topical options like podophyllin, imiquimod cream, trichloroacetic acid and cryotherapy, injectable options like interferon and 5-fluoroucil, and surgical options like excision, fulguration, cryotherapy, and laser removal. However, the treatment is usually short-lived, and the patients are subjected to multiple repeat procedures because of high recurrence and low clearance rates. Surgical management has the highest clearance rate. There are several surgical modalities including excision, electrosurgical fulguration (ESF), and LASER vaporization. LASER techniques work directly to destroy/transect the lesion, cause necrosis of infected keratinocytes and induce local inflammation. LASER treatment is also reported to have minimal local surrounding tissue injury and sphincter injury, and less pain and discomfort. For this reason, LASER therapy has been increasingly used to remove anogenital warts, and is a standard of care treatment of condyloma. We hypothesize that LASER vaporization is effective to treat perianal condyloma and may have clinical benefits over ESF. We will compare postoperative outcomes such as pain, healing, cosmesis and recurrence following either treatment method.

ELIGIBILITY:
Inclusion Criteria: Adults (>18) treated in our CRS department for perianal condyloma, not previously treated surgically, English speaking patients.

Exclusion Criteria: <18, intra-anal condyloma, previously treated for condyloma, other skin diseases in the perianal region, limited English proficiency.

* Adults unable to consent- exclude
* Individuals who are not yet adults (infants, children, teenagers)- exclude
* Pregnant women- exclude
* Prisoners- exclude

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Anal Condyloma | 6 months
  Comparison of recurrence of anal condyloma within 6 months among LASER group and ESF group.

SECONDARY OUTCOMES:
Comparison of Postoperative Pain and associated outcomes | 6 months
  Comparison of postoperative outcomes among LASER group and ESF group. The outcomes of interest are postoperative pain, healing time, and cosmesis.
Incidence of Treatment-Emergent complications | 6 months
  Major complications including soft tissue infection and hemorrhage.